CLINICAL TRIAL: NCT07220070
Title: Communication Compass Feedback
Brief Title: Communication Compass
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-00752
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Patient Education and Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Group A) (Experimental): Participants assigned to Group A receive algorithm-based feedback reports plus standard curriculum.
  Interventions: Other: Algorithm-Based Feedback Reports; Other: Standard Curriculum
- Control Group (Group B - Delayed Exposure) (Active Comparator): Participants assigned to Group B receive the standard curriculum with usual summary reports. Group members also receive algorithm-based feedback after study completion).
  Interventions: Other: Standard Curriculum

INTERVENTIONS:
Other: Algorithm-Based Feedback Reports — Feedback reports that provide personalized, near-real-time feedback on internal medicine residents' patient education and counseling (PEC) communication skills.
  Arms: Intervention Group (Group A)
Other: Standard Curriculum — Standard summary reports on internal medicine residents' patient education and counseling (PEC) communication skills.

SUMMARY:
The primary purpose of this study is to develop, implement, and validate algorithm-based feedback reports (Communication Compass) that provides personalized, near-real-time feedback on internal medicine residents' patient education and counseling (PEC) communication skills. This research aims to address critical gaps in current communication skills training by leveraging technology to enhance the frequency and specificity of communication skills feedback while maintaining ethical standards and established educational effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Post-graduate year 1 (PGY1) and post-graduate year 2 (PGY2) internal medicine residents enrolled in NYU Langone Health residency programs.
* Medical school graduates enrolled in ACGME-accredited internal medicine residency programs
* Residents who routinely participate in required educational activities including OSCEs and clinical assessments

Exclusion Criteria:

• Individuals who do not meet the criteria established in the 'Inclusion Criteria.'

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-27 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Resident Competency | Up to Year 2
  Percentage of residents rated "well done" on PEC items across all PGY2 Objective Structured Clinical Examination (OSCE) cases.
Resident Improvement | Up to Year 1, Up to Year 2
  Percentage of residents showing PEC rating improvement from PGY1 to PGY2 OSCE.

CONTACTS AND LOCATIONS:
Overall Officials: Yuliya Yoncheva, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Non-federal sponsor.